CLINICAL TRIAL: NCT06337773
Title: Developing the Precision Nursing Education Program Through the E-flipped Classroom Model to Improve the Quality of Life Among Young Colorectal Cancer Survivors
Brief Title: Developing the Precision Nursing Education Program to Young Colorectal Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-BR-112-036
Record Dates: First submitted 2024-03-17; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: depression; young colorectal cancer survivors; precision nursing education
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The survivors receiving 8 weeks (90 mins per weeks) on-line percious nursing education intervention
  Interventions: Behavioral: 8-weeks's on-line precision nursing education program
- Control group (No Intervention): As usual

INTERVENTIONS:
Behavioral: 8-weeks's on-line precision nursing education program — The intervention involved 8-weeks's on-line precision nursing education program, including Qigong exercise, and mindfulness training.
  Arms: Treatment group

SUMMARY:
This study is aimed to demonstrate the long-term effectiveness of 8-week precision nursing education program through the e-flipped classroom model for YCC survivors and provide a compliant strategy to improve quality of life and emotional status of these patients.

DETAILED DESCRIPTION:
Background: In recent years, there has been an increase in case number of patients with young colon cancer (YCC). After curative treatment, YCC survivors have more opportunities to meet physical, social and economic burdens. Furthermore, YCC survivors may suffer poor quality of life and depression symptoms related to disease treatments and specific post-treatment care intervention is in unmet need.

Objective: The precision nursing education program will be developed through the eflipped classroom model, including the care of physical symptom based on the patients' needs, Qigong exercise, and mindfulness training. To evaluate the effect of these interventions, the questionnaire of the quality of life of YCC survivors will be employed.

Method: A randomized controlled trial containing 110 patients aged between 20 and 50 years old will be conducted. After completion of curative operation and adjuvant treatments, the subjects will be randomly assigned to a control group, in which routine nursing education care will be provided, and an intervention group, in which 8-week precision nursing education program through the e-flipped classroom model will be applied. The outcome measures include EORTC QLQ-C30, EORTC QLQ-CR29, BDI Depression Scale, Constructed Meaning Scale and FFMQ. The time-points of outcome measures include pre-intervention, post-intervention (at the end of the intervention), and 3, 6 and 9 months after the end of intervention. Univariate analyses will be performed to examine the intervention outcomes among basic characteristics of subjects. Correlation analyses will be performed to investigate the relationships between intervention outcomes and different variables. Comparisons of mean scores in the dependent variables between the experimental group and control group over the five time-points will be used in the generalization of estimating equation models.

Contribution: This study is aimed to demonstrate the long-term effectiveness of 8- week precision nursing education program through the e-flipped classroom model for YCC survivors and provide a compliant strategy to improve quality of life and emotional status of these patients.

ELIGIBILITY:
Inclusion Criteria:

* survivor was diagnosed as colon, rectal, colorectal, or/and anal cancer
* aged at least 20 years
* have had completed cancer treatments within the five years prior to enrolling in the study.
* agree and obtain written consent
* could using the online media(ex: Zoom or Google meet..) to attend intervention course

Exclusion Criteria:

* diagnosed with stage IV cancer
* had a recurrence of CRC cancer
* had the other type cancer diagnosis
* now are undering cancer treatment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
The depression symptoms on young colorectal cancer survivors | Baseline (T0) and then week 8 (the end of the intervention) (T1), the 3rd month (T2), the 6th month (T3), and the 9th month (T4).
  The 21-item Beck Depression Inventory-II (BDI-II) is using to measure the depression syptoms. It comprised of 21 items. The total score range of BDI-II was from 0 to 63, with higher scores indicating greater severity of depression. The BDI-II cutoff point for clinical depression is a total score of >13.

SECONDARY OUTCOMES:
Dispositional mindfulness status on young colorectal cancer survivors | Baseline (T0) and then week 8 (the end of the intervention) (T1), the 3rd month (T2), the 6th month (T3), and the 9th month (T4).
  The 39-item Five Facet Mindfulness Questionnaire24 measures dispositional mindfulness including observing, describing, acting of awareness, nonjudging, and nonreactivity to inner experience. Participants indicated their responses on a 5-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), with higher scores indicating higher levels of dispositional mindfulness. The Cronbach's alpha for the full scale in this study was 0.87.
General quality of life on young colorectal cancer survivors | Baseline (T0) and then week 8 (the end of the intervention) (T1), the 3rd month (T2), the 6th month (T3), and the 9th month (T4).
  General quality of life are measuring by the EORTC QLQ-C30. EORCT QLQ-C30 measures CRC patients' general physical status that consisted including functions and symptoms status. The ranges of these two scales were from 0 to 100, with higher scores indicating the higher levels of function status and symptoms distress.
Colorectal specific quality of life on young colorectal cancer survivors | Baseline (T0) and then week 8 (the end of the intervention) (T1), the 3rd month (T2), the 6th month (T3), and the 9th month (T4).
  Colorectal specific quality of life are measuring by the QLQ- CR29. EORTC QLQ-CR29 measures CRC patients' colorectal functions and symptoms.The ranges of these two scales were from 0 to 100, with higher scores indicating the higher levels of function status and symptoms distress.
Cancer threat appraisal on young colorectal cancer survivors | Baseline (T0) and then week 8 (the end of the intervention) (T1), the 3rd month (T2), the 6th month (T3), and the 9th month (T4).
  Constructed Meaning Scale (CMS)15 measures participants' cancer threat appraisal. The CMS relies on eight items to measure patients' perceptions with respect to identifying CRC, their interpersonal re- lationships, and their future lives. The ratings are made on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with lower scores indicating a more negative cancer meaning status and appraisal of CRC as a greater threat.

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.